CLINICAL TRIAL: NCT04161079
Title: Evaluation of the 5-Year Safety and Performance of the Medtentia Annuloplasty Ring in Adults - Follow-Up to Clinical Investigation 2010-040
Brief Title: 5-Year Follow-Up Safety and Performance Evaluation of the Medtentia Annuloplasty Ring in Adults
Status: Completed | Type: Observational
Sponsor: Medtentia International Ltd Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-040FU5
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency
Keywords: Mitral valve; Mitral surgery; Mitral repair; Mitral annuloplasty; Mitral valve surgery; Mitral valve repair; Mitral valve annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAR population: Subjects, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040
  Interventions: Device: Medtentia Annuloplasty Ring (MAR)

INTERVENTIONS:
Device: Medtentia Annuloplasty Ring (MAR) — Mitral valve repair using the MAR performed in clinical investigation 2010-040

SUMMARY:
Single-center clinical investigation is to evaluate long-term safety and performance of the Medtentia Annuloplasty Ring (MAR) in 11 patients who underwent successful mitral valve (MV) surgery using Medtentia's MAR system in clinical investigation 2010-040 performed during June 2011 - April 2016.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Subject had a successful MAR implantation in clinical investigation 2010-040.
* Subject is willing to participate in the follow-up study and to comply with the requirements of the Clinical Investigation Plan.

Exclusion Criteria:

* Subjects who participated in the clinical investigation 2010-040 but had the MAR replaced with another mitral valve repair ring or system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects, who underwent mitral valve repair operation with successful MAR implantation in clinical investigation 2010-040.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapio Aalto, MD, Principal Investigator — Mehiläinen hospital
Locations (1):
- Mehiläinen hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medtentia Company Webpage — http://medtentia.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each MAR patient attended a single visit at the investigational site Mehiläinen hospital, Helsinki, during the period from 08 Nov 2019 to 29 Jan 2020. Maximum of 11 MAR patients who underwent successful MAR implantation and completed 2010-040 clinical investigation were anticipated to be qualifying for this follow-up clinical investigation.
Pre-assignment Details: This follow up investigation compared 5-year timepoint data with the 2-year results of 2010-040 investigation, therefore enrollment numbers differ in the Protocol Section (7) and in the Participant Flow (12).
  7 MAR patients returned for 2010-040FU5 follow-up visit and 3 of these were with MAR Classic, 1 with MAR Regular and 3 with MAR Expanded.
Groups:
- MAR Population: Subjects, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040
  For some of outcome measures it is defined as MAR Population >5 Years Follow-up Timepoint
Period: Clinical Investigation 2010-040
Arm/Group | MAR Population
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1
Period: 2010-040FU5 >5 Years Follow-up
Arm/Group | MAR Population
Started (It is follow-up group from the clinical investigation 2010-040.) | 7 (Of 11 subjects 3 refused to participate and 1 died.)
Completed | 7 (Timepoint distribution for individual patients ranged approximately 6-8 yrs after MAR implantation.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MAR Population: Baseline data was presented for this follow-up clinical investigation 2010-040FU5 population (7 participants) which included participants who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040 and were enrolled in this follow-up clinical investigation 2010-040FU5.
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040.
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Finland | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety: the Occurrence, Nature and Frequency of Significant Medical Events
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Number; unit: Events
Groups:
- MAR Population: 2010-040FU5 >5 years follow-up population
  Subjects, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Events | 0

2. Primary Outcome: Performance: Change in Mitral Regurgitation (MR) as Measured by Trans-Thoracic Echocardiography (TTE)
Description: Success will be defined as no change or any improvement in MR class as described in the American College of Cardiology/ American Heart Association (ACC/AHA) Guidelines
Time Frame: from 2-year follow-up data point to more than 5 years post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Investigation 2010-040 2-year Follow-up: Data for MAR population during clinical Investigation 2010-040, collected 2 years after MAR implantation
- 2010-040FU5 >5 Years Follow-up: Subjects, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040
Arm/Group | Clinical Investigation 2010-040 2-year Follow-up | 2010-040FU5 >5 Years Follow-up
Number analyzed (Participants) | 11 | 7
Participants
  I - None/Trivial | 8 | 5
  II - Mild | 3 | 2
  III - Moderate | 0 | 0
  IV - Severe | 0 | 0

3. Secondary Outcome: Safety: All-Cause Mortality
Description: Collected retrospectively
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Population: All-cause mortality data was collected retrospectively since the last visit of clinical investigation 2010-040. During the course of the recruitment it became known that one MAR patient had died and it accounted for 9% of all-cause mortality rate in all 11 MAR patients. The cause of death was noncardiac-related and was not attributed to MAR.
Measure: Count of Participants; unit: Participants
Groups:
- MAR Population: Clinical investigation 2010-040 2-year follow-up population
  Subjects, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040
Arm/Group | MAR Population
Number analyzed (Participants) | 11
Participants | 1

4. Secondary Outcome: Safety: the Occurrence, Nature and Frequency of Adverse Device Effects (ADEs) and/or Device Deficiencies
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Number; unit: Events
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Events | 0

5. Secondary Outcome: Safety: Number of Cardiovascular Admissions
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Number; unit: Cardiovascular Admissions
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Cardiovascular Admissions | 0

6. Secondary Outcome: Safety: the Number of Subjects With Clinically Significant Abnormal Findings
Description: The number of subjects with clinically significant abnormal findings in TTE, electrocardiography (ECG), or vital signs and type of abnormal findings will be listed and tabulated
Time Frame: day of study visit
Measure: Count of Participants; unit: Participants
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Participants | 0

7. Secondary Outcome: Performance: Change in Mitral Regurgitation Parameters (Left Ventricle Reverse Remodeling), as Measured by TTE
Description: Change from the clinical investigation 2010-040 2-year follow-up in the following MR parameters, as measured by TTE:
  - Left ventricle reverse remodeling: left ventricular inner dimension systole and diastole (the dimension of inner edge to inner edge, perpendicular to the long axis of the left ventricle, at the level of the mitral valve leaflet tips, measured at end-systole and end-diastole)
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Clinical Investigation 2010-040 2-year Follow-up | 2010-040FU5 >5 Years Follow-up
Number analyzed (Participants) | 11 | 7
millimeters
  Left Ventricular Inner Dimension Systole | 38 [36 to 43] | 41 [39 to 47]
  Left Ventricular Inner Dimension Diastole | 51 [49 to 52] | 56 [51 to 59]

8. Secondary Outcome: Performance: Changes in New York Heart Association (NYHA) Classification When Compared to the Clinical Investigation 2010-040 2-year Follow-Up Visit
Description: Defined as assessment of NYHA functional class status at clinical Investigation 2010-040 2-year follow-up visit and at this investigation visit more than 5 years post-procedure
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Investigation 2010-040 2-year Follow-up | 2010-040FU5 >5 Years Follow-up
Number analyzed (Participants) | 11 | 7
Participants
  Class I | 11 | 1
  Class II | 0 | 6
  Class III | 0 | 0
  Class IV | 0 | 0

9. Secondary Outcome: Performance: Number of Subjects With Recurrence of Mitral Regurgitation
Description: Recurrence of mitral regurgitation is defined as changing of mitral regurgitation to moderate or severe according to ACC/AHA classification determined by TTE
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Participants | 0

10. Other Pre Specified Outcome: Number of Subjects With Re-operation or Mitral Valve Reintervention Due MAR Performance Failure or Malfunction
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Participants | 0

11. Other Pre Specified Outcome: Quality of Life Scores as Measured by the 15D© Questionnaire
Description: 15D© questionnaire investigates the standard of quality of life (QOL15D) through a general health assessment and not specific to a particular disease or age. It is a 15-domain (mobility, vision, hearing, breathing, sleeping, eating, speech, excretion, usual activities, mental function, discomfort and symptoms, depression, distress, vitality and sexual activity) questionnaire. Each domain score ranges from 1 (no problems) to 5 (extreme problems), with lower scores reflecting better health-related functional status.
Time Frame: day of study visit
Population: Response for quality of life scores for sexual activity domain of 15D© questionnaire received from 6 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | MAR Population
Number analyzed (Participants) | 7
Participants
  QOL15D-Mobility: 1 | 5
  QOL15D-Mobility: 2 | 2
  QOL15D-Mobility: 3 | 0
  QOL15D-Mobility: 4 | 0
  QOL15D-Mobility: 5 | 0
  QOL15D-Vision: 1 | 5
  QOL15D-Vision: 2 | 2
  QOL15D-Vision: 3 | 0
  QOL15D-Vision: 4 | 0
  QOL15D-Vision: 5 | 0
  QOL15D-Hearing: 1 | 5
  QOL15D-Hearing: 2 | 2
  QOL15D-Hearing: 3 | 0
  QOL15D-Hearing: 4 | 0
  QOL15D-Hearing: 5 | 0
  QOL15D-Breathing: 1 | 3
  QOL15D-Breathing: 2 | 4
  QOL15D-Breathing: 3 | 0
  QOL15D-Breathing: 4 | 0
  QOL15D-Breathing: 5 | 0
  QOL15D-Sleeping: 1 | 5
  QOL15D-Sleeping: 2 | 1
  QOL15D-Sleeping: 3 | 1
  QOL15D-Sleeping: 4 | 0
  QOL15D-Sleeping: 5 | 0
  QOL15D-Eating: 1 | 7
  QOL15D-Eating: 2 | 0
  QOL15D-Eating: 3 | 0
  QOL15D-Eating: 4 | 0
  QOL15D-Eating: 5 | 0
  QOL15D-Speech: 1 | 6
  QOL15D-Speech: 2 | 1
  QOL15D-Speech: 3 | 0
  QOL15D-Speech: 4 | 0
  QOL15D-Speech: 5 | 0
  QOL15D-Excretion: 1 | 6
  QOL15D-Excretion: 2 | 1
  QOL15D-Excretion: 3 | 0
  QOL15D-Excretion: 4 | 0
  QOL15D-Excretion: 5 | 0
  QOL15D-Usual activities: 1 | 4
  QOL15D-Usual activities: 2 | 3
  QOL15D-Usual activities: 3 | 0
  QOL15D-Usual activities: 4 | 0
  QOL15D-Usual activities: 5 | 0
  QOL15D-Mental function: 1 | 3
  QOL15D-Mental function: 2 | 4
  QOL15D-Mental function: 3 | 0
  QOL15D-Mental function: 4 | 0
  QOL15D-Mental function: 5 | 0
  QOL15D-Discomfort and symptoms: 1 | 4
  QOL15D-Discomfort and symptoms: 2 | 3
  QOL15D-Discomfort and symptoms: 3 | 0
  QOL15D-Discomfort and symptoms: 4 | 0
  QOL15D-Discomfort and symptoms: 5 | 0
  QOL15D-Depression: 1 | 4
  QOL15D-Depression: 2 | 3
  QOL15D-Depression: 3 | 0
  QOL15D-Depression: 4 | 0
  QOL15D-Depression: 5 | 0
  QOL15D-Distress: 1 | 4
  QOL15D-Distress: 2 | 3
  QOL15D-Distress: 3 | 0
  QOL15D-Distress: 4 | 0
  QOL15D-Distress: 5 | 0
  QOL15D-Vitality: 1 | 2
  QOL15D-Vitality: 2 | 5
  QOL15D-Vitality: 3 | 0
  QOL15D-Vitality: 4 | 0
  QOL15D-Vitality: 5 | 0
  QOL15D-Sexual activity: number analyzed (Participants) | 6
  QOL15D-Sexual activity: 1 | 3
  QOL15D-Sexual activity: 2 | 3
  QOL15D-Sexual activity: 3 | 0
  QOL15D-Sexual activity: 4 | 0
  QOL15D-Sexual activity: 5 | 0

12. Secondary Outcome: Performance: Change in Mitral Regurgitation Parameters (Coaptation Height), as Measured by TTE
Description: Change from the clinical investigation 2010-040 2-year follow-up in the coaptation height, as measured by TTE
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Population: At clinical investigation 2010-040 2-year follow-up timepoint data was available for 9 of 11 participants.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Clinical Investigation 2010-040 2-year Follow-up | 2010-040FU5 >5 Years Follow-up
Number analyzed (Participants) | 9 | 7
millimeters | 7.4 (2.3) | 3.9 (5.4)

ADVERSE EVENTS:
Time Frame: since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure
Description: The occurrence, nature and frequency of adverse device effects (ADEs) and/or device deficiencies (DDs) since the last visit of clinical investigation 2010-040.
  Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for the Clinical Investigation 2010-040 2-year Follow-up group, therefore total number of participants at risk is "0".
Groups:
- Clinical Investigation 2010-040 2-year Follow-up: Data for MAR population during clinical Investigation 2010-040, 11 participants, collected for the time frame since the last visit of clinical investigation 2010-040 to more than 5 years post-procedure (2010-040FU5)
  Serious adverse events and other adverse events data collected only for study 2010-040FU5 participants
- 2010-040FU5 >5 Years Follow-up: Patient, who underwent MV repair operation with successful MAR implantation in clinical investigation 2010-040 and were enrolled in clinical investigation 2010-040FU5
  Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the MAR performed in clinical investigation 2010-040
Arm/Group | Clinical Investigation 2010-040 2-year Follow-up | 2010-040FU5 >5 Years Follow-up
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/7

LIMITATIONS AND CAVEATS:
The investigation was limited by its retrospective nature and design. Due to small study sample not all the comparisons of the parameters at the two timepoints (2-year and 5-year follow-up) could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04161079/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT04161079/SAP_001.pdf